CLINICAL TRIAL: NCT05260775
Title: Intelligent Evaluation and Supervision of Cataract Surgery
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, principal investigator, Sun Yat-sen University
Other Study IDs: CS-2022
Record Dates: First submitted 2022-02-27; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Cataract
Keywords: cataract surgery
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Development Dataset: 12 cataract surgery steps including(1) main incision formation, (2) side incision formation, (3) ophthalmic viscoelastic device (OVD) injection, (4) capsulorrhexis formation, (5) hydrodissection, (6) phaco, (7) cortical material removal, (8) intraocular lens (IOL) implantation, (9) OVD removal, (10) IOL centration and (11) wound closure through corneal hydration, and (12) idle phases.
  Interventions: Other: Evaluation test: cataract surgery steps
- Validation Dataset: 12 cataract surgery steps including(1) main incision formation, (2) side incision formation, (3) ophthalmic viscoelastic device (OVD) injection, (4) capsulorrhexis formation, (5) hydrodissection, (6) phaco, (7) cortical material removal, (8) intraocular lens (IOL) implantation, (9) OVD removal, (10) IOL centration and (11) wound closure through corneal hydration, and (12) idle phases.
  Interventions: Other: Evaluation test: cataract surgery steps
- Test Dataset: 12 cataract surgery steps including(1) main incision formation, (2) side incision formation, (3) ophthalmic viscoelastic device (OVD) injection, (4) capsulorrhexis formation, (5) hydrodissection, (6) phaco, (7) cortical material removal, (8) intraocular lens (IOL) implantation, (9) OVD removal, (10) IOL centration and (11) wound closure through corneal hydration, and (12) idle phases.
  Interventions: Other: Evaluation test: cataract surgery steps

INTERVENTIONS:
Other: Evaluation test: cataract surgery steps — The development datasets were used to train the deep learning model. The validation and test group were used to optimize hyperparameters

SUMMARY:
Research purpose: intelligent identification and evaluation of cataract surgery steps Research methods: A total of 9 items (such as gender, age, visual acuity, etc.) were extracted from the surgical videos of senile cataract patients and the clinical data recorded by the electronic medical record system. The machine learning algorithm 3D-CNN was applied to identify the 11 steps in cataract surgery and the pictures (blank pictures) without instrument manipulation on the eyeball during the operation. Six key cataract surgery steps were scored using deep learning algorithms (probability smoothing window and softmax). We employ precision, precision, recall, and F1-score to evaluate the model's performance for recognizing surgical steps. To evaluate the reliability of the model's scoring of surgical steps, we used a human-machine comparison method to calculate the agreement (kappa value) between machine and expert scores.

ELIGIBILITY:
Inclusion Criteria:

-Videos of phacoemulsification and IOL implantation for senile cataracts will be included

Exclusion Criteria:

-The peak signal-to-noise ratio (PSNR) is utilized to assess whether a video was blurred. If the PSNR of a video was less than 20 decibels (dBs), the whole video was discarded.

Ages: 50 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants who had senile cataracts and phacoemulsification and IOL implantation in the Zhongshan Ophthalmic Centre (ZOC, Guangzhou, Guangdong, China) and Shenzhen Eye Hospital (Shenzhen, Guangdong, China)
Sampling Method: Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Accuracy | baseline
  The investigators will calculate accuracy of deep learning system and compare this index between deep learning system and human doctors

SECONDARY OUTCOMES:
kappa | baseline
  Cohen's kappa coefficient was calculated to assess the agreement between the grades given by human doctors and DeepSurgery

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, M.D., Ph.D., Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China